CLINICAL TRIAL: NCT04001387
Title: Feasibility of Real-time Ultrasound-guided Spinal Anesthesia Using Dynamic Needle Tip Positioning
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Tae Kyong Kim, Assistant Professor, Seoul National University Hospital
Other Study IDs: 20-2019-32
Record Dates: First submitted 2019-06-26; First posted 2019-06-28 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Regional Anesthesia Morbidity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spinal anesthesia
  Interventions: Procedure: Real-time ultrasound guided spinal anesthesia

INTERVENTIONS:
Procedure: Real-time ultrasound guided spinal anesthesia — The neuraxial US scan will be performed with the patient in the lateral position with the hip and knees flexed using full aseptic technique. The spinal needle will be inserted in real-time under direct ultrasound guidance using dynamic needle tip positioning to administer the spinal anesthetic.

SUMMARY:
Confirming the L4-L5 or L3-L4 vertebrae level with ultrasound in real time for adults who scheduled elective surgery under spinal anesthesia, and introduce the spinal needle into the subarachnoid space. The ultrasound probe continues to track needle tips in real time by sliding/tilting with short axis view. Check that the spinal needle reaches subarachnoid space, and that CSF is released through the needle hub, and administer the drug.

In this process, it is recorded by observing the success of the procedure, the time taken for each step, the number of needle position changes, NRS pain score of the subject, satisfaction with anesthesia, and its side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients who scheduled for elective surgery under spinal anesthesia
* Age >= 20

Exclusion Criteria:

* Patient refusal
* Coagulopathy (INR ≥1.2, anticoagulant therapy)
* Sepsis or local infection at the site of injection
* BMI > 35
* Spine deformity

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who scheduled for elective surgery under spinal anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-10-27 (Estimated); Primary Completion 2020-05-26 (Estimated); Study Completion 2020-06-26 (Estimated)

PRIMARY OUTCOMES:
Successful perfomance of spinal anesthesia | Assessed at time of spinal anesthetic injection (baseline)
  Rate of successful performance of real-time ultrasound guided spinal needle insertion using dynamic needle tip positioning

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grau T, Leipold RW, Conradi R, Martin E, Motsch J. Ultrasound imaging facilitates localization of the epidural space during combined spinal and epidural anesthesia. Reg Anesth Pain Med. 2001 Jan-Feb;26(1):64-7. doi: 10.1053/rapm.2001.19633. No abstract available. PMID 11172514
- [Background] Kil HK, Cho JE, Kim WO, Koo BN, Han SW, Kim JY. Prepuncture ultrasound-measured distance: an accurate reflection of epidural depth in infants and small children. Reg Anesth Pain Med. 2007 Mar-Apr;32(2):102-6. doi: 10.1016/j.rapm.2006.10.005. PMID 17350519
- [Background] Carvalho JC. Ultrasound-facilitated epidurals and spinals in obstetrics. Anesthesiol Clin. 2008 Mar;26(1):145-58, vii-viii. doi: 10.1016/j.anclin.2007.11.007. PMID 18319185
- [Background] Grau T, Leipold RW, Fatehi S, Martin E, Motsch J. Real-time ultrasonic observation of combined spinal-epidural anaesthesia. Eur J Anaesthesiol. 2004 Jan;21(1):25-31. doi: 10.1017/s026502150400105x. PMID 14768920
- [Background] Hanada S, Van Winkle MT, Subramani S, Ueda K. Dynamic ultrasound-guided short-axis needle tip navigation technique vs. landmark technique for difficult saphenous vein access in children: a randomised study. Anaesthesia. 2017 Dec;72(12):1508-1515. doi: 10.1111/anae.14082. Epub 2017 Oct 6. PMID 28983903
- [Background] Kiberenge RK, Ueda K, Rosauer B. Ultrasound-Guided Dynamic Needle Tip Positioning Technique Versus Palpation Technique for Radial Arterial Cannulation in Adult Surgical Patients: A Randomized Controlled Trial. Anesth Analg. 2018 Jan;126(1):120-126. doi: 10.1213/ANE.0000000000002261. PMID 29135593
- [Background] Liu L, Tan Y, Li S, Tian J. "Modified Dynamic Needle Tip Positioning" Short-Axis, Out-of-Plane, Ultrasound-Guided Radial Artery Cannulation in Neonates: A Randomized Controlled Trial. Anesth Analg. 2019 Jul;129(1):178-183. doi: 10.1213/ANE.0000000000003445. PMID 29787409
- [Background] Takeshita J, Yoshida T, Nakajima Y, Nakayama Y, Nishiyama K, Ito Y, Shimizu Y, Takeuchi M, Shime N. Dynamic Needle Tip Positioning for Ultrasound-Guided Arterial Catheterization in Infants and Small Children With Deep Arteries: A Randomized Controlled Trial. J Cardiothorac Vasc Anesth. 2019 Jul;33(7):1919-1925. doi: 10.1053/j.jvca.2018.12.002. Epub 2018 Dec 4. PMID 30638922